CLINICAL TRIAL: NCT03004196
Title: Comparison of Efficacy Of Probiotic Toothpaste and Chlorhexidine Mouthwash To Reduce Streptococcus Mutans in Plaque Around Orthodontic Brackets
Brief Title: Comparison of Efficacy Of Probiotic Toothpaste and Chlorhexidine Mouthwash To Reduce S.Mutans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peoples University, Bhanpur, Bhopal (Other)
Responsible Party: Principal Investigator, Chandrika Dubey, Post-Graduate Student, Peoples University, Bhanpur, Bhopal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CD-01
Record Dates: First submitted 2016-12-02; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: White Spot Lesion of Tooth; Long Term Adverse Effects; Caries, Dental; Orthodontic Appliance Complication
Keywords: White Spot Lesion; Probiotics; Chlorhexidine; Streptococcus Mutans; Fixed Orthodontic Treatment
MeSH Terms: conditions — Long Term Adverse Effects; Dental Caries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Active Comparator): They were not given probiotic toothpaste or chlorhexidine mouthwash
  Interventions: Other: Control Group
- Probiotic Group (Experimental): Patients were asked to brush twice daily with given "G.D Probiotic Toothpaste" and were asked not to eat or drink anything for half-an-hour.
  Interventions: Drug: Probiotic Toothpaste
- Chlorhexidine Mouthwash Group (Experimental): Patients were asked to rinse daily with "Dr. Reddy's Clohex" chlorhexidine mouthwash of 10ml without dilution for three times a day after meals (Breakfast, Lunch Dinner) for 3-4 minutes and were asked not to eat or drink anything for half-an-hour.
  Interventions: Drug: Dr. Reddy's Clohex

INTERVENTIONS:
Drug: Probiotic Toothpaste — G.D Probiotic Toothpaste bacteriocin Lactic Acid Bacteria
  Other Names: G.D Probiotic Toothpaste
  Arms: Probiotic Group
Drug: Dr. Reddy's Clohex — 0.20% Chlorhexidine Mouthwash
  Other Names: Chlorhexidine Mouthwash
  Arms: Chlorhexidine Mouthwash Group
Other: Control Group — No Probiotic toothpaste & Chlorhexidine Mouthwash
  Arms: Control Group

SUMMARY:
Orthodontic appliance causes increase in plaque accumulation, especially around brackets, wires and attachments. Advances in orthodontics in recent time have led to improved quality of appliance and treatment procedures ultimately resulting in improvised standard of patient care.

These bacteria metabolize different kind of carbohydrates accumulated around orthodontic appliances and create acidic environment in the oral cavity leading to enamel demineralization around the brackets and white spot lesions.

This study was carried out to evaluate and compare the efficacy of probiotic toothpaste and chlorhexidine mouthwash in patients undergoing orthodontic treatment with individuals who are not using them.

DETAILED DESCRIPTION:
INTRODUCTION - When the basic oral hygiene is poor, orthodontic appliances create areas where plaque gets accumulated, especially around brackets, bands, wires, and other attachments; this facilitates the development of white spot lesions. Probiotics act by competitively inhibiting the pathogenic bacteria because they have greater adhesion to the tissues while Chlorhexidine is often used as an active ingredient in mouthwash designed to reduce dental plaque around orthodontic appliances. AIM & OBJECTIVE - The objectives of the study is to evaluate and compare the effects of the topical application of probiotic toothpaste and chlorhexidine mouthwash on the Streptococcus Mutans levels in the plaque of orthodontic patients hence improving the oral micro-flora of oral cavity by competitive inhibition of Streptococcus Mutans in plaque present around brackets.

MATERIAL & METHOD - The study consists of thirty randomly selected orthodontic patients undergoing fixed appliance treatment. The patients were divided into three groups - Control Group (Group 1), Probiotic Toothpaste Group (Group 2) & Chlorhexidine Mouthwash Group (Group 3). Samples were collected at two times interval: before the study began (Phase 1) and after thirty days (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic Treatment With The Straight Wire Appliance (MBT, 0.022-in Slot; 3M Unitek, Monro- Via, Calif), Permanent Dentition (Excluding Third Molars)
* Good General Health (No Significant Medical History Or Drug Use During The Last Month)
* No Anti-inflammatory Or Antibiotic Medications Taken In The Month Before The Study
* No Chewing Gum Or, Mouthwash Used In The Last Week And During The Study
* Habit Of Brushing Twice Daily With Fluoride Toothpaste

Exclusion Criteria:

-Patient with poor periodontal condition Patient with known medical condition e.g. Subacute bacterial, endocarditis , diabetes, valvular disease ,anaemia etc

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Control Group/Probiotic Toothpaste/Chlorhexidine Mouthwash | 1 Month
  Probiotic Toothpaste & Chlorhexidine Mouthwash Reduced S.mutans when compared to Control Group

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Chandrika Dubey, MDS, Principal Investigator — Peoples University
Locations (1):
- Peoples College Of Dental Science & Research Center, Bhopal, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jose JE, Padmanabhan S, Chitharanjan AB. Systemic consumption of probiotic curd and use of probiotic toothpaste to reduce Streptococcus mutans in plaque around orthodontic brackets. Am J Orthod Dentofacial Orthop. 2013 Jul;144(1):67-72. doi: 10.1016/j.ajodo.2013.02.023. PMID 23810047